CLINICAL TRIAL: NCT04299841
Title: Stress Disorder Post-stroke: Observational Study of the Evaluation of Post Traumatic Stress Post Stroke (Stroke Post Traumatic Disorder)
Brief Title: Observational Study of the Evaluation of Post Traumatic Stress Post Stroke
Acronym: SPTD
Status: Withdrawn | Type: Observational
Why Stopped: lack of time
Sponsor: Ch Mont de Marsan (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A01962-55
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PCL 5; Stroke
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective, observational, multicentre study evaluates the existence of Post-traumatic stress disorder following a stroke at 3 and 6 months after the management of the patient.

Questionnaires will be used to assess the presence of stroke post traumatic disorder.

The evaluation of stroke post traumatic disorder would allow to underline the importance of the awareness of the care teams in the the screening of these disorders and to evaluate if the Post-traumatic Stress Disorder Checklist Scale (PCL5) is an effective screening tool.

ELIGIBILITY:
Inclusion Criteria:

* Patient age > 18years old
* Patient registered with a social security scheme
* Patient who was given a written information and who gave his/her non-opposition
* Patient who was hospitalized with a diagnosis of stroke in the neurology department and oriented to the post-stroke consultation (3 months after the hospital discharge) or un the follow-up care and readaptation department of hospital center of Dax or Mont de Marsan

Exclusion Criteria:

* Patient with a serious disability sequelae (mRS>3),
* Patient without enough level of proficiency in the French language,
* Patient with neurocognitive and neurocognitive disorder diagnosed,
* Patient with history of significant psychiatric disorders diagnosed,
* Patient with seve aphasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient who was hospitalized with a diagnosis of stroke in the neurology department and oriented to the post-stroke consultation (3 months after the hospital discharge) or un the follow-up care and readaptation department of hospital center of Dax or Mont de Marsan
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the number of patients managed for stroke and presenting Stroke Post Traumatic Disorder at 3 months after stroke | at time of inclusion (3 months after stroke)
  Evaluate the number of patients managed for stroke and presenting Stroke Post Traumatic Disorder at 3 months after stroke. This evaluation will be made by completion of PCL-5 questionnaire (Post-traumatic stress disorder checklist version DSM-5 (DSM:Diagnostic and Statistical Manuel of Mental Disorders)). A PCL-5 positive score will be an indicator of post-traumatic stress disorder correlated with stroke.

SECONDARY OUTCOMES:
Evaluate the number of patients managed for stroke and presenting Stroke Post Traumatic Disorder at 3 and at 6 months | at time of inclusion (3 months after stroke) and 6 months after stroke (study participation duration for patient: 3 months)
  Evaluate the number of patients managed for stroke and presenting Stroke Post Traumatic Disorder at 3 and at 6 months. This evaluation will be made by completion of PCL-5 questionnaire (Post-traumatic stress disorder checklist version DSM-5). A PCL-5 positive score will be an indicator of post-traumatic stress disorder correlated with stroke. Two timepoint: 3 months and 6 months after stroke.
Evaluate the number of patients presenting a depressive state at 3 months | at time of inclusion (3 months after stroke)
  Evaluate the number of patients presenting a depressive state at 3 months after stroke. This evaluation was done by completion of HAD (Hospital Anxiety and Depression scale) questionnaire. A score between 8 and 10 will identify a doubtful depressive symptomatology and a score Superior to 11 will identify a certain depressive symptomatology.
Evaluate the number of patients under antidepressant or anxiolytics treatment before the stroke | at time of inclusion (3 months after stroke)
  The evaluation of the number of patients under antidepressant or anxiolytics treatment before the stroke will be made by the collection of previous treatments of the patient.
Evaluate the PCL-5 questionnaire as a screening tool of the stroke post traumatic disorder | at time of inclusion (3 months after stroke) and 6 months after stroke (study participation duration for patient: 3 months)
  Evaluate the PCL-5 questionnaire as a screening tool of the stroke post traumatic disorder by completion of PCL-5 questionnaire at two timepoint (3 and 6 months post-stroke). The presence of Post-traumatic Stress Disorder will be defined by threshold value of 38 as the total score on the PCL-5 questionnaire.
Evaluate the traumatic history of the patient before the occurrence of the stroke | at time of inclusion (3 months after stroke)
  Evaluate the number of patients presenting a depressive state at 3 months after stroke. This evaluation was done by completion of Trauma History Questionnaire (THQ).
Evaluate the existence of a peritraumatic dissociation at the time of the occurrence of the stroke | at time of inclusion (3 months after stroke)
  Evaluate the number of patients presenting a depressive state at 3 months after stroke. This evaluation was done by completion of PDEQ (Peritraumatic Dissociative Experience Questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Harold PERDIGNON, Principal Investigator — CH de Dax; Francine CLEMENTI, MD, Study Director — CH de Dax
Locations (1):
- centre hospitalier Dax, Dax, France